CLINICAL TRIAL: NCT06901804
Title: Effect of Pilates Core Stabilization in Adjunct With Plyometric Shoulder Training on Low Back Pain in Fast Bowlers: a Randomized Controlled Trial
Brief Title: Effect of Pilates Core Stabilization in Adjunct With Plyometric Shoulder Training on Low Back Pain in Fast Bowlers(RCT)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MSRSW/Batch-Fall23/777
Record Dates: First submitted 2025-03-23; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Control Groups; Physical Therapy Modalities; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental)
  Interventions: Diagnostic Test: Experimental Group (training and stabilization)
- Control Group (Active Comparator)
  Interventions: Combination Product: Control Group (physiotherapy and exercise)

INTERVENTIONS:
Diagnostic Test: Experimental Group (training and stabilization) — Plyometric Shoulder Training [28] and Pilates Core Stabilization [27]
  Exercise 1-2 weeks (rep × kg) 3-4 weeks (rep × kg) 5-6 weeks (rep × kg) Throwing Movements Medicine ball chest pass 8 × 1 kg 10 × 2 kg 12 × 3 kg Medicine ball step and pass 8 × 1 kg 10 × 2 kg 12 × 3 kg Medicine ball side throw 8 × 1 kg 10 × 2 kg 12 × 3 kg Tubing Plyos IR/ER 8 × 10 10 × 10 12 × 12 Tubing Plyos Diagonal 8 × 10 10 × 10 12 × 12 Tubing Plyos Biceps 8 × 10 10 × 10 12 × 12 Plyo Push-ups (boxes) 8 × 10 10 × 10 12 × 12 Push-ups (clappers) 8 × 10 10 × 10 12 × 12
  Arms: Experimental Group
Combination Product: Control Group (physiotherapy and exercise) — Physiotherapy Care for Low Back Pain [30] Exercise Week 1-2 (Sets x Reps/Duration) Week 3-4 (Sets x Reps/Duration) Week 5-6 (Sets x Reps/Duration) Plank 3 x 20 sec 3 x 30 sec 4 x 45 sec Bicycle Crunches 3 x 12 3 x 15 4 x 20-25 Leg Raises 3 x 12 3 x 15 4 x 20-25 Russian Twists 3 x 20 3 x 25 4 x 30-35 Slump Exercise 3 x 10 3 x 12 4 x 15-18 Bridge Exercise with Swiss Ball 3 x 12 3 x 15 4 x 18
  Arms: Control Group

SUMMARY:
This RCT will seek to determine both the Pilates core stabilization and plyometric shoulder training on LBP in fast bowlers. The research problem will emphasize the absence of detailed rehabilitation protocols that address the upper and lower limb strength dysfunction, pain, quality of life, and biomechanics of fast bowlers. Prior literature has not examined the combined use of these two training interventions to address LBP, which affects the performance of fast bowlers. In this study, participants will be randomly assigned to two groups. Group A (experimental) will receive Pilates core stabilization and plyometric shoulder training, while Group B (control) will receive conventional physiotherapy for LBP. There will be two sessions per week for six weeks, and the intensity of the exercises will gradually increase to address athletes' strength, flexibility, and movement control.

DETAILED DESCRIPTION:
Assessments will be conducted using multiple scales of upper limb strength for the Cricket Ball Throw Test, lower limb strength for the Vertical Jump Test, Quality of Life for the Oswestry Disability Index, biomechanics analysis to determine movement efficiency and Pain Intensity for Numeric Pain Rating Scale. This study will give information about the efficiency of adding core and shoulder training to managing LBP in fast bowlers, increasing their athletic performance and bringing helpful value to the sports and physiotherapy domain.

ELIGIBILITY:
Inclusion Criteria:

* Age between 17-25 years
* Male cricket players
* Playing cricket for more than 2 years
* Low back pain without radiation
* Chronic low back pain for more than 3 months
* Non-specific mechanical type without identifiable specific anatomical or neurophysiological causative factors and medically fit

Exclusion Criteria:

* Any pathological condition of the spine, hip, knee, and pelvis.
* Any history of musculoskeletal injury in the past 6 months.
* Any history of a neurological condition.
* Uncontrolled metabolic disorders such as Diabetes Mellitus
* Any surgical h/o shoulder or elbow in the past 6 months

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
NPRS (Numeric Pain Rating Scale) | 12 Months
  The NPRS denotes pain severity on a whole-number scale, ranging from 0 to 10, with 0 meaning no pain at all and 10 signifying the worst pain one has ever experienced. A lower score on the scale indicates a reduced level of pain as perceived by the patients having ICC 0.95.
CBTT (Cricket Ball Throw Test) | 12 months
  This test evaluates upper limb strength and coordination by documenting the distance a cricket ball attained (in meters). More separation suggests better strength of the upper limbs and better place and movement of the limbs with ICC: 0.92.
VJT (Vertical Jump Test) | 12 months
  The VJT quantifies lower limb explosive power by only assessing the vertical jump height expressed in centimeters. Higher values denote better control of the lower extremities with ICC 0.95.

CONTACTS AND LOCATIONS:
Locations (1):
- Pakistan Cricket Board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No